CLINICAL TRIAL: NCT02506309
Title: Prospective Randomized Comparison of the Trans-obturator Mid-urethral Sling and the Single-incision Sling in Women With Stress Urinary Incontinence
Brief Title: Trans-obturator Mid-urethral Sling and the Single-incision Sling in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Martin Huser, professor, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrnoUH
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIS single incision sling (Experimental): SIS - Innovative fixation single incision sling A third generation of the Mid-urethral slings inserted through a SIS single incision sling (SIS) to treat female stress urinary incontinence (SUI).
  Interventions: Device: SIS - Innovative fixation single incision sling
- TOT trans obturator tape/sling (Active Comparator): TOT - inside-out trans-obturator tape/sling Trans-obturator slings (TOT) now represent a gold standard in the treatment of female stress urinary incontinence (SUI).
  Interventions: Device: TOT - inside-out trans-obturator tape/sling

INTERVENTIONS:
Device: TOT - inside-out trans-obturator tape/sling — Patients were randomized by envelope technique at the time of surgery indication to either TOT or SIS anti-incontinence surgical procedure with mid-urethral slings (MUS)
  Other Names: Gynecare TVT Obturator System (Ethicon)
  Arms: TOT trans obturator tape/sling
Device: SIS - Innovative fixation single incision sling — Patients were randomized by envelope technique at the time of surgery indication to either TOT or SIS anti-incontinence surgical procedure with mid-urethral slings (MUS)
  Other Names: Ophira (Promedon)
  Arms: SIS single incision sling

SUMMARY:
Mid-urethral slings (MUS) now represent a gold standard in the treatment of female stress urinary incontinence (SUI). Second generation trans-obturator slings (TOT) have proven to be as effective as retropubic tension-free vaginal tape (TVT) with fewer major complications. A third generation of the MUS inserted through a single vaginal incision (SIS) has become a means to overcome significant post-operative groin pain. Novel types of SIS with a more robust and adjustable anchoring mechanism can assure adequate long-lasting attachment to the obturator membrane (OM). Objective of this study was to compare an inside-out TOT with an innovative fixation SIS in randomized controlled trial on patients undergoing their primary surgery for urodynamic SUI.

DETAILED DESCRIPTION:
Objective of this study was to compare an inside-out TOT (Gynecare TVT Obturator System, Ethicon) with an innovative fixation SIS (Ophira, Promedon) in randomized controlled trial on patients undergoing their primary surgery for urodynamic SUI.

A prospective randomized controlled trial (RCT) is performed in one tertiary referral urogynecology center from January 2015 thru December 2015. Study included women with pure or predominant urodynamic SUI confirmed during cystometry by positive standardized cough stress test (CST) with urinary bladder filling of 250 ml in lithotomy position. Study was carried out on a Caucasian Czech (central European) population. A study power analysis was calculated with an expected objective cure rate of minimum 80 % for both patient groups, false non-match rate (alpha) of 0.05, and false match rate (beta) of 0.10. A minimum sample size of 80 patients was required for each group.

ELIGIBILITY:
Inclusion Criteria:

Women with pure or predominant urodynamic stress urinary incontinence confirmed during filling cystometry by positive standardized cough stress test (CST) with urinary bladder filling of 250 ml in lithotomy position.

Exclusion Criteria:

* patients with predominant urge incontinence
* patients with intrinsic sphincter deficiency (MUCP<20 cmH2O)
* pelvic organ prolapse (POP-Q>2)
* previous urinary incontinence surgery
* previous pelvic organ prolapse surgery
* presence of other pelvic organ pathology.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

REFERENCES:
- [Background] Ogah J, Cody DJ, Rogerson L. Minimally invasive synthetic suburethral sling operations for stress urinary incontinence in women: a short version Cochrane review. Neurourol Urodyn. 2011 Mar;30(3):284-91. doi: 10.1002/nau.20980. PMID 21412819
- [Background] Nambiar A, Cody JD, Jeffery ST. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2014 Jun 1;(6):CD008709. doi: 10.1002/14651858.CD008709.pub2. PMID 24880654
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839
- [Derived] Huser M, Hudecek R, Belkov I, Horvath I, Jarkovsky J, Tvarozek S. Safety and Efficacy of Single Incision Sling Versus Midurethral Sling in the Treatment of Stress Urinary Incontinence: A Randomized Controlled Trial. Urogynecology (Phila). 2023 Feb 1;29(2):113-120. doi: 10.1097/SPV.0000000000001284. PMID 36735422

RESULTS

PARTICIPANT FLOW:
Groups:
- TOT Trans Obturato Tape/Sling: TOT - inside-out trans-obturator tape/sling Trans-obturator slings (TOT) now represent a gold standard in the treatment of female stress urinary incontinence (SUI).
  TOT - inside-out trans-obturator tape/sling: Patients were randomized by envelope technique at the time of surgery indication to either TOT or SIS anti-incontinence surgical procedure with mid-urethral slings (MUS)
Period: Overall Study
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Started | 84 | 84
Completed | 66 | 64
Not Completed | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.6) | 62.3 (10.3) | 63.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 168
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Negative Cough Stress Test (CST)
Description: Negative cough stress test four years after incontinence surgery.
Time Frame: four years
Measure: Number; unit: percentage of participants
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Number analyzed (Participants) | 66 | 64
percentage of participants | 86.4 | 83.1

2. Primary Outcome: Patient Global Impression of Improvement (PGI-I) Score
Description: Patient Global Impression of Improvement (PGI-I) score four years after incontinence surgery. The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale). It is a simple, direct, easy to use scale that is intuitively understandable to clinicians
  1. Very much better
  2. Much better
  3. A little better
  4. No change
  5. A little worse
  6. Much worse
  7. Very much worse
Time Frame: four years
Measure: Mean (Full Range); unit: units on PGI-I scale
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Number analyzed (Participants) | 66 | 64
units on PGI-I scale | 1.4 [0 to 7] | 1.3 [0 to 7]

3. Secondary Outcome: Number of Participants With Major Perioperative Complications
Time Frame: one month
Measure: Number; unit: participants
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Number analyzed (Participants) | 84 | 84
participants | 0 | 0

4. Secondary Outcome: Number of Participants With Major Postoperative Complications
Time Frame: four years
Measure: Number; unit: participants
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Number analyzed (Participants) | 66 | 64
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | SIS Single Incision Sling | TOT Trans Obturato Tape/Sling
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/64
Other Adverse Events (participants affected / at risk) | 0/66 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes